CLINICAL TRIAL: NCT06702514
Title: Effectiveness of Balneotherapy in the Treatment of Hand Osteoarthritis: a Randomized Controlled Trial
Brief Title: Balneotherapy in Hand Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, Ass. Prof., Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SABALNEO
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Hand Osteoarthritis
MeSH Terms: interventions — Exercise; Paraffin; Balneology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balneotherapy Group (Experimental): This group will receive 20 minutes of paraffin and 20 minutes of balneotherapy on both hands, five times a week for 4 weeks, for a total of 20 sessions, using one session per day. In addition, a daily exercise program (15 minutes of joint range of motion, 15 minutes of strengthening exercises) will be given once a day, accompanied by a physiotherapist.
  Interventions: Other: Exercise; Other: Paraffin; Other: Balneotherapy
- Control Group (Active Comparator): The control group was planned to receive 20 minutes of paraffin treatment on both hands, five times a week for 4 weeks, one session per day for a total of 20 sessions. In addition, a daily exercise program (15 minutes of joint range of motion, 15 minutes of strengthening exercises) will be given once a day, accompanied by a physiotherapist.
  Interventions: Other: Exercise; Other: Paraffin

INTERVENTIONS:
Other: Exercise — After their treatment, both groups will be given a daily exercise program (15 minutes of range of motion, 15 minutes of strengthening exercises) once a day, accompanied by a physiotherapist.
Other: Paraffin — It was planned to apply paraffin treatment to both hands for 20 minutes, five times a week for 4 weeks, using one session per day for a total of 20 sessions.
Other: Balneotherapy — The balneotherapy group will receive 20 minutes of paraffin and 20 minutes of balneotherapy on both hands, five times a week for 4 weeks, one session per day for a total of 20 sessions. The spa treatment will be given in the form of a 20-minute full body bath in the pool in each session. The spa water temperature will be 38-40 degrees Celsius.
  Arms: Balneotherapy Group

SUMMARY:
There are a limited number of studies in the literature on the effectiveness of balneotherapy in hand osteoarthritis. The aim of this study was to evaluate the effects of balneotherapy on pain, manual skills, functionality and quality of life in patients with hand osteoarthritis who have undergone balneotherapy.

DETAILED DESCRIPTION:
Hand osteoarthritis (OA) is a chronic and disabling disease that can cause pain and functional limitations. The estimated radiological prevalence of hand OA is approximately 54-67% in the adult population aged 55 years and older. This prevalence is expected to increase as the number of elderly people increases. Current guidelines strongly recommend exercise as a nonpharmacological approach to the treatment of hand osteoarthritis, while thermal treatments and paraffin therapy are conditionally recommended.

Balneotherapy is defined as a natural mineral water bath and is one of the most widely used nonpharmacological complementary treatments for different rheumatic diseases in many European countries, Turkey, Israel and Japan. In the last decade, related advances have made it possible to understand the therapeutic effects of balneotherapy in some musculoskeletal disorders.

The effectiveness is achieved through a combination of mechanical, thermal and chemical effects. Warm stimuli increase the pain threshold and provide analgesia in nerve endings. The EULAR task force's recommendation for hand OA, which suggests local heat application (e.g. paraffin wax, hot pack) as a useful treatment, also draws attention to the effect of heat. Spa treatment triggers a series of neuroendocrine reactions and particularly induces the release of adrenocorticotropic hormone (ACTH), cortisol, prolactin and growth hormone (GH).

Thermomineral water baths have a small effect on pain, a moderate effect on symptoms related to other musculoskeletal diseases and up to 3 months of pain relief; it is considered to be more beneficial than tap water or no treatment for the improvement of symptoms related to musculoskeletal diseases. Even a single balneotherapy procedure can provide pain relief.

There are a limited number of studies in the literature on the effectiveness of balneotherapy in hand osteoarthritis. The aim of this study was to evaluate the effects of balneotherapy on pain, manual skills, functionality and quality of life in patients with hand osteoarthritis who have undergone balneotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50-75
* Hand osteoarthritis diagnosed according to ACR criteria

Exclusion Criteria:

* Non-cooperative patients
* Trauma or surgery to the hand region in the last 6 months
* Infection
* Infection, loss of sensation, metal implant in the treatment area
* Injection to the hand joints in the last 3 months
* Physical therapy and rehabilitation to the hand region in the last 3 months
* Balneotherapy in the last 3 months
* Inflammatory rheumatic diseases
* NSAI use
* Planning pregnancy during pregnancy or treatment
* Malignancy
* Presence of a neurological disease
* Hand-wrist entrapment neuropathy
* Loss of muscle strength or sensation in the hand
* Uncontrolled cardiopulmonary disease
* Open wound
* Orthopedic condition that would prevent entering the spa

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual Pain Scale (VAS) | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  VAS which is easy to understand, apply and interpret, and provides valid and reliable data in a short time, is the most commonly used method in clinics. With a 100 mm visual linear scale, the patient is told that there is no pain at point 0, and that the most severe pain they have ever felt at point 100, and the patient is asked to put a mark on the point corresponding to their pain.
Palm-to-finger distance | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  Palm-to-finger distance Used to assess hand joint mobility. Obtained by measuring the distance (in millimeters) between the fingertip of the second to fifth finger and the distal palmar crease while making a full fist and adding the distances (higher scores indicate greater limitations).
The Australian / Canadian Osteoarthritis Hand Index (AUSCAN) | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  It was developed specifically for use in hand osteoarthritis. It is recommended for use in clinical studies by OMERACT (Outcome Measures in Rheumatology Clinical Trials Group). It evaluates hand functions, pain and stiffness in patients with hand osteoarthritis. It consists of three subscales: Hand pain (5 items), hand stiffness (1 item), hand function (9 items). A 5-point Likert scale (0=none, 4=severe) LK 3.0 is used. Its validity and reliability have been demonstrated in osteoarthritis.
Hand Osteoarthritis Functional Index | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  It is a 10-question questionnaire. Answers are scored on a 4-point scale: 0 = Possible without difficulty; 1 = Possible with some difficulty; 2 = Possible with great difficulty; 3 = Impossible. The total score for the questionnaire ranges from 0 to 30. A higher score indicates a more severe functional limitation. Validity and reliability in Turkish have been demonstrated.
Jamar Dynamometer | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  Measurements will be made by sitting with the shoulder adducted and neutrally rotated, adjacent to the body, elbow 90 degrees flexed, wrist 0-30 degrees dorsiflexed and 0-15 degrees ulnar deviation, thumb up. Measurements will be repeated three times with 5-second intervals on the affected hand and the average of the three measurements will be recorded in kilograms. Finger grip strength will be assessed with the 'Jamar digital pinchmeter'. Patients will be placed in a sitting position with the wrist 90° flexed and the forearm in a neutral position. Measurements will be made bilaterally in three different positions as lateral, palmar and fingertip grips. Patients will be asked to squeeze with maximum force and each measurement will be taken three times and the average will be recorded in kg.

SECONDARY OUTCOMES:
Nine Hole Pag Test | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  This test measures manual dexterity based on performance (seconds). A wooden board with nine holes on it, 9 short wooden sticks and a box in which the wooden sticks can be placed are placed in front of the patient. The patient is asked to place the wooden sticks in the box into the holes on the board as quickly as possible using the hand to be evaluated, then is asked to put the sticks back into the box one by one. The test completion time is determined by a stopwatch
Jebsen Taylor Hand Function Test | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  Test items are turning cards, picking up small objects and throwing them into a tin can, stacking backgammon tiles, writing, jumping 5 light tin cans across, jumping 5 heavy tin cans across, collecting 5 dried kidney beans using a dessert spoon The test materials include detailed instructions for use in the test manual. In order to ensure a standard arrangement of the objects used, a scaled board and a stopwatch are included in the test materials to measure the time the activities are performed. Before the test is administered, the person is shown how to do it. Explaining that the test is performed against time is necessary for the patient's motivation. The patient starts with the start command and the stopwatch is stopped when the activity is completed.
Health Assessment Questionnaire (HAQ) | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  HAQ was developed for the assessment of patients with rheumatic diseases. It consists of 20 questions related to eight activities (items); dressing, getting up, eating, walking, hygiene, grasping and activities of daily living are questioned. HAQ reflects the functional status of patients and this questionnaire has been shown to correlate with disease activity markers. Each item or question is rated on a scale of 0 to 3, with 0 (normal/no difficulty), 1 (some difficulty), 2 (much difficulty), and 3 (unable to do). The 8 category scores are averaged, which represent an overall score from 0 (no disability) to 3 (completely disabled).
  Scores 0-1 indicates mild to moderate disability, 1-2 indicates moderate to severe disability, and 2-3 indicates severe to very severe disability.
SF-36 Quality of Life Scale | Before treatment (T0), after treatment (4. week) (T1), 8. week (T2)
  SF-36 is a generic quality of life scale. It is evaluated between 0-100 points. It was created to evaluate health status. It contains a total of 36 items. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.There is a Turkish validity and reliability study.

IPD SHARING:
Plan to Share IPD: No